CLINICAL TRIAL: NCT07010042
Title: Effects of Preoperative Anxiety and Preemptive Analgesia on Postoperative Delirium in Septo/Rhinoplasty Surgery
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, medical doctor, Zonguldak Bulent Ecevit University
Other Study IDs: 2020Septo/Rhinoplasty Surgery
Record Dates: First submitted 2025-05-23; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Preoperative Anxiety; Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Bays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group P: n: 43patients: Group P: Patients administered iv 1 gr paracetamol 30 minutes before surgery
  Interventions: Other: The Beck Anxiety Inventory (BAI) of adult patients
- Group K:n:43 patients: Group K: Patients administered iv 1 gr paracetamol 15 minutes before the end of surgery
  Interventions: Other: The Beck Anxiety Inventory (BAI) of adult patients

INTERVENTIONS:
Other: The Beck Anxiety Inventory (BAI) of adult patients — Postoperative 0,5,10,15 minutes , RSAS and NRS values
  Other Names: Postoperative agitation in adult patients is assessed with the Riker Sedation-Agitation Scale (RSAS).; The Numerical Pain Scale (NRS) is used to evaluate postoperative pain in adult patients.

SUMMARY:
Effects of Preoperative Anxiety and Preemptive Analgesia on Postoperative Delirium in Septo/Rhinoplasty Surgery

DETAILED DESCRIPTION:
It is known that preoperative anxiety causes postoperative agitation.

In adult patients, preoperative anxiety is assessed with the Beck Anxiety Inventory (BAI) and BAI≥16 is considered 'anxious'. Postoperative agitation is assessed with the Riker Sedation-Agitation Scale (RSAS) and RSAS ≥5 is considered agitated, pain is assessed with the Numerical Pain Scale (NRS) >4 is considered postoperative pain. Measurements were recorded at 0, 5, 10 and 15 minutes postoperatively.

There are factors such as inhalation agents, preoperative anxiety and postoperative pain in its etiology.

ELIGIBILITY:
Inclusion Criteria:

* - 18-65 years old,
* ASA I-II risk group
* Those who will be operated under general anesthesia under elective conditions.
* Will undergo surgery for Septo/Rhinoplasty
* Patients whose informed consent form was read to their parents was obtained

Exclusion Criteria:

* -Those do not want to participate in the study,
* ASA III -IV-V patients
* Having a history of drug allergy and drug interaction,
* Having a history of systemic disease such as heart, kidney, liver failure,
* Having a history of bleeding diathesis,
* Difficult intubation expected,
* Obese,
* Emergency patients,
* Mental-motor retarded,
* Having psychiatric and neurological diseases,
* Those with chronic drug use

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 86
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Effects of Preoperative Anxiety and Preemptive Analgesia on Postoperative Delirium in Septo/Rhinoplasty Surgery | During the first 15 minutes postoperatively
  The correlation between the BAI values of the groups and the RSAS scores and NRS values Beck Anxiety Scale Scoring 8-15 points are categorized as mild anxiety symptoms, 2. 16-25 points are moderate anxiety symptoms, 3. 26-63 points are severe anxiety symptoms.
  Riker Sedation-Agitation Scale:
  7-Dangerous agitation 6-Very agitated 5-Agitated 4-Calm and cooperative 3-Sedated 2-Very sedated
  1-Unarousable Numerical Rating Scale Scores range from 0-10, with higher scores indicating greater pain intensity.
Preemptive Analgesia for Postoperative Agitation in Septo/Rhinoplasty Surgery | During the first 15 minutes postoperatively
  The relationship between the BAI values of the groups and the RSAS scores and NRS The correlation between the BAI values of the groups and the RSAS scores and NRS values Beck Anxiety Scale Scoring 8-15 points are categorized as mild anxiety symptoms, 2. 16-25 points are moderate anxiety symptoms, 3. 26-63 points are severe anxiety symptoms. Riker Sedation-Agitation Scale: 7-Dangerous agitation 6-Very agitated 5-Agitated 4-Calm and cooperative 3-Sedated 2-Very sedated 1-Unarousable Numerical Rating Scale Scores range from 0-10, with higher scores indicating greater pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided